CLINICAL TRIAL: NCT03945032
Title: Digital Technology for Parents in Pediatric Oncology: Development and Implementation
Brief Title: TICOP Mobile App and E-platform: Providing Information and Support for Parents Caring for Their Child Cancer Survivor
Acronym: TICOP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: In process (technical improvements)
Sponsor: Vander Haegen Marie (Other)
Responsible Party: Sponsor-Investigator, Vander Haegen Marie, Doctor of Psychology (Ph.D) (Uliège), University of Liege
Organization: University of Liege (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1819-30 (Uliège)
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Mobile Application
Keywords: Parent of a childhood cancer survivor; E-platform; TICOP mobile App

STUDY DESIGN:
Intervention Model Description: 8 parents of a childhood cancer survivor will participate in this study (baseline + three times per year). Parents will answer on the TICOP mobile app. Parents will pretest the "TICOP" mobile app. One year later, they will return to the laboratory in order to brainstorm with the principal investigator (an accredited psychologist) about the mobile App and its operation and usefulness.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 8 parents of a childhood cancer survivor (Experimental): Parent moves the cursor by analogy on their mobile phone (as a visual anagogic scale) four times per year (baseline; month 4; month 8 and month 12).
  Interventions: Other: TICOP

INTERVENTIONS:
Other: TICOP — Parent moves the cursor by analogy on their mobile phone (as a visual anagogic scale) four times per year (baseline; month 4; month 8 and month 12).

SUMMARY:
This study aims to develop a mobile App (named "TICOP") for parents of a childhood cancer survivor and an E-Platform for health professionals which work in pediatric oncology area.

The core objective is to evaluate the effects of these two digital tools (mobile app and platform) in the detection and prevention among parents of a childhood cancer survivor.

DETAILED DESCRIPTION:
Parents of a childhood cancer survivor face ongoing social, and psychological challenges that may result in enduring illness and caregiving related distress and vulnerabilities. It has been described namely: post posttraumatic stress symptoms [PTSS], lingering worries, anxiety and depression. While strategies and interventions to minimize the child's distress have become part of comprehensive medical care in paediatrics, it also becomes urgent to develop research into parents of a childhood cancer survivor in order to: [1] train the medical staff to identify the serious issue of parental distress ; [2] detect other markers of vulnerabilities (e.g. pessimism, anxiety trait) and [3] provide them with a personalized psychological intervention. This would allow vigilance of the medical staff in detecting parents' distress and could defuse their descent into a vicious circle of psychosocial difficulties.

Up to now, empirical findings suggest the importance to develop a screening tool for parents of a CCS in order to detect any parent who presents several difficulties and to propose personal intervention. To the investigator's knowledge, there is no tool to detect and prevent psychological distress among parents of a childhood cancer survivor.

The TICOP mobile app consists of seven axis of evaluation and detection for parents of a childhood cancer survivor:

Parent moves the cursor by analogy on their mobile phone (as a visual anagogic scale) four times per year (baseline; month 4; month 8 and month 12).

Axis 1: sociodemographic (e.g. gender, marital status) (14 items) Axis 2: psychosomatic symptoms (insomnia, migraine) (16 items) Axis 3: psychological symptoms (e.g. depression, anxiety) (13 items) Axis 4: parental needs (e.g. social support, information) (9 items) Axis 5: parental resources (e.g. emotional support) (8 items) Axis 6: parental risk factors (e.g. anxiety, intolerant of uncertainty) (5 items) Axis 7: parental protective factors (e.g. optimistic,extraverted) (6 items)

All information will be automatically sent in real time into the E-platform. This digital tool allows to obtain a parental state follow-up for the health professional (e.g. oncologist, psycho-oncologist).

ELIGIBILITY:
Inclusion Criteria:

* Parent of a childhood cancer survivor (mother and father)
* Child who had been diagnosed in remission since 1 years until 10 years (without relapse)
* Neoadjuvant chemotherapy during treatments
* Fluency in French speaking
* No previous evidence of mental illness.

Exclusion Criteria:

* Diagnosis of cancer treated only by surgery or radiotherapy (with no adjuvant chemotherapy)
* Benign tumor
* Child has a relapse or died
* Non-French-speaking parents
* previous evidence of mental illness.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Psychological symptoms (created for the needs of the study) | Measure assessing change between four time points (change from Baseline at 4 months, 8 months and 12 months)
  13 items ranged between 0% at 100% [Visual Analog Scale] Scale range : 0 = rarely; 1 = occasionally ; 2 = often; 3 = mostly
  Note. Results are significant when the score is above 25% for one single item with at least two occurrences over time period.
Psychosomatic symptoms (created for the needs of the study) | Measure assessing change between four time points (change from Baseline at 4 months, 8 months and 12 months)
  16 items ranged between 0% at 100% [Visual Analog Scale] Scale range : 0 = rarely; 1 = occasionally ; 2 = often; 3 = mostly
  Note. Results are significant when the score is above 25% for one single item with at least two occurrences over time period.
Parental needs (created for the needs of the study) | Measure assessing change between four time points (change from Baseline at 4 months, 8 months and 12 months)
  9 items ranged between 0% at 100% [Visual Analog Scale]
Parental resources (created for the needs of the study) | Measure assessing change between four time points (change from Baseline at 4 months, 8 months and 12 months)
  8 items ranged between 0% at 100% [Visual Analog Scale]
Parental risk factors (created for the needs of the study) | Measure assessing change between four time points (change from Baseline at 4 months, 8 months and 12 months)
  5 paired-items ranged between 0% at 100% [Visual Analog Scale]
  Note. Results are significant when the score is above 25% for one single item with at least two occurrences over time period.
Parental protective factors (created for the needs of the study) | Measure assessing change between four time points (change from Baseline at 4 months, 8 months and 12 months)
  6 paired-items ranged between 0% at 100% [Visual Analog Scale]
  Note. Results are significant when the score is above 25% for one single item with at least two occurrences over time period.
Sociodemographic questionnaire (parents of a childhood cancer survivor) (created for the needs of the study) | Baseline
  14 items (multiple-choice response)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Vander Haegen, Dr., Principal Investigator — University of Liege
Locations (1):
- University of Liège (Unit: Health Psychology), Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vander Haegen M, Etienne AM. Intolerance of uncertainty in parents of childhood cancer survivors: A clinical profile analysis. J Psychosoc Oncol. 2018 Nov-Dec;36(6):717-733. doi: 10.1080/07347332.2018.1499692. Epub 2018 Nov 14. PMID 30427278
- [Background] Vander Haegen M, Etienne AM. Intolerance of uncertainty as the vulnerability factor among parents of childhood cancer survivors: A 3-month follow-up study. J Psychosoc Oncol. 2018 Jul-Aug;36(4):437-453. doi: 10.1080/07347332.2018.1443192. Epub 2018 May 14. PMID 29757114
- [Background] Vander Haegen M, Luminet O. Stress, Psychosocial Mediators, and Cognitive Mediators in Parents of Child Cancer Patients and Cancer Survivors: Attention and Working Memory Pathway Perspectives. J Psychosoc Oncol. 2015;33(5):504-50. doi: 10.1080/07347332.2015.1067279. PMID 26181302